CLINICAL TRIAL: NCT00123877
Title: Phase II, Open Label, Non-Randomized, Efficacy and Safety Study of an Intravenous Formulation of the Anthracycline Analog, GPX-100, in the Treatment of Metastatic Breast Cancer
Brief Title: Study of GPX-100 in the Treatment of Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gem Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPX-100-003
Record Dates: First submitted 2005-07-23; First posted 2005-07-26 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Breast Cancer; Metastasis
Keywords: Breast; Cancer; Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms

INTERVENTIONS:
Drug: GPX-100 (13-deoxydoxorubicin)

SUMMARY:
The purpose of this early Phase II multicenter trial is to determine the objective clinical response to GPX-100, an anthracycline similar to doxorubicin, in up to 40 patients with newly diagnosed metastatic breast cancer. GPX-100 is unique among anthracyclines because it is not converted to doxorubicinol during metabolism in the body. This metabolite has been shown to be a major cause of damage to the heart (cardiotoxicity) in laboratory studies. Eligible patients who are enrolled in this study will receive GPX-100 as a single agent at the beginning of as many as 8 three week long cycles of chemotherapy. Objective measurements of tumor response will be made by computed tomography (CT) scans.

DETAILED DESCRIPTION:
Study Design - Two-stage, multicenter, open-label, non-randomized study with intravenous (IV) dose administration of GPX-100 and limited dose-escalation and de-escalation. After confirmation of the maximum tolerated dose (MTD) and interim analysis of efficacy and safety (Stage I), if necessary the study cohort will be enlarged to confirm the estimate of clinical efficacy (Stage II) using the established MTD.

Sample Size - 20 patients in Stage I and up to 20 patients in Stage II.

Dosage Form - IV solution of sterilized lyophilized powder in Sodium Chloride (NaCl) for Injection, USP (0.9%).

Doses - 140 mg/m2 GPX-100 with escalation to 170 mg/m2 and de-escalation to 105 mg/m2 depending upon clinical response and toxicity.

Administration - One IV infusion every 3 weeks for up to 8 doses.

Efficacy Parameters - Activity of GPX-100 will be evaluated in terms of measurable tumor response and disease progression according to RECIST criteria. Blood samples will be obtained for determination of pharmacokinetic parameters and the presence of doxorubicinol following the first dose of GPX-100.

Safety Parameters - Dose tolerance and treatment toxicity, especially cardiotoxicity, of GPX-100 will be evaluated. A baseline medical history including Karnofsky Performance Status and a physical examination, hematology profile (CBC, differential, platelet count), chemistry profile including electrolytes, serum calcium, liver and renal function tests, urinalysis, chest and abdominal CT scans, and a bone scan will be done. Interval history with adverse event (AE) assessment and performance status, physical examination, and hematology and clinical chemistry profile will be repeated every 3 weeks during treatment. In addition, hematology and chemistry profiles will be repeated weekly between treatment visits. Chest and abdominal CTs and bone scans will be repeated at 6-week intervals as appropriate for tumor assessment. An MRI of the brain will be performed at the baseline visit if clinically indicated. Urinalysis will be repeated at six-week intervals during treatment. Cardiotoxicity will be assessed with ECG and MUGA scans at baseline, every 6 weeks during treatment, and 6-8 weeks after the last dose of GPX-100. There will be continued follow-up at 6-8 week intervals if indicated by changing cardiac function until normal or stable. Treatment will be discontinued if there is objective disease progression or unacceptable treatment toxicity. A follow-up visit will occur 6-8 weeks after the last treatment visit for each patient, whether the study was completed per protocol or the patient discontinues study treatment early for any reason. The following evaluations will be performed at the follow-up visit: physical examination, adverse event assessment, ECG, MUGA scan, hematology and clinical chemistry profiles, and urinalysis. Serum pregnancy tests will be performed at baseline and at the follow-up visit, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patient is female and at least 18 years of age.
* Patient has histologically or cytologically confirmed diagnosis of breast cancer and clinical or pathologic evidence of metastatic disease at the time of presentation or following remission that resulted from standard therapy, which may have included adjuvant chemotherapy and hormonal therapy.
* Patient has at least one measurable soft tissue metastatic lesion excluding bone metastases, brain metastases, ascites, and pleural effusions. A measurable lesion must be present on a radiographic study (CT scan is preferred) and must be > 20 mm maximum diameter on plain film or traditional CT scan (> 10 mm on spiral CT).
* Patient has progressive disease based on the appearance of new lesions or an increase of at least 25% in the diameter of measurable lesions.
* Patient has a performance status of at least 70% on Karnofsky scale; patient has a predicted life expectancy of at least 24 weeks.
* Patient has not received any investigational agents within 4 weeks of this study and no chemotherapy for metastatic or recurrent disease. Patients should receive supportive care as indicated. Patients requiring palliative radiation therapy should receive their course of radiation treatment before entering the study.
* Patient may have received adjuvant chemotherapy provided that the patient's relapse has occurred at least 12 months subsequent to completion of adjuvant therapy.
* Patient may have received unlimited prior hormonal therapy, provided that it was completed at least 4 weeks prior to the first study treatment and there is radiographic evidence of progression following hormonal withdrawal.
* Patient has fully recovered from any previous surgery (at least 4 weeks since major surgery) and radiation therapy (at least 4 weeks since treatment).
* Patient has recovered from reversible toxicity from prior therapy. Permanent and stable side effects or changes are acceptable.
* Patient has adequate hematological function, including neutrophils > 2,000 cells/uL, platelets > 100,000/uL, and hemoglobin > 10.0 gm/dL.
* Patient has adequate organ function defined as a bilirubin within the normal range; AST < 1.5 times the upper limit of normal (ULN; < 2.5 times the ULN with liver involvement); alkaline phosphatase < 1.5 times ULN (< 3 times the ULN with liver involvement, or < 5 times the ULN with bone but no liver involvement); and serum creatinine < 2.0 mg/dL.
* Patient has a normal ejection fraction (by institutional criteria) as determined by resting MUGA scan.
* Patient has a negative pregnancy test prior to study entry if premenopausal or if less than 12 months after menopause. Premenopausal patients must use a medically effective form of contraception during the treatment period.
* Patient is willing and able to comply with all study protocol requirements. The patient or a legally authorized representative must fully understand all elements of the informed consent and have signed the informed consent according to institutional and federal regulatory requirements.

Exclusion Criteria:

* Patient is male.
* Patient is pregnant or breast-feeding.
* Patient has a history of hypersensitivity to anthracyclines.
* Patient has received a cumulative dose of doxorubicin that exceeds 300 mg/m2 or a cumulative dose of epirubicin that exceeds 540 mg/m2.
* Patient has received an anthracycline or other chemotherapy as adjuvant treatment for breast cancer within 12 months prior to entry into the study.
* Patient has received an anthracycline or other chemotherapy regimen for metastatic or recurrent disease. Anthracycline-based adjuvant chemotherapy for initial disease does not exclude enrollment.
* Patient has metastases involving the central nervous system (CNS).
* Patient has metastases limited to bone.
* Prior history of congestive heart failure (CHF), myocardial infarction within 6 months prior to enrollment, active ischemic heart disease, or uncontrolled hypertension.
* Patient requires active medical therapy for CHF or arrhythmia.
* Patient has participated in a study of any investigational drug within 4 weeks prior to the first study treatment.
* Patient has a history within the past 5 years of other prior primary malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or another cancer from which the patient has been disease-free for at least 5 years.
* Patient has received chemotherapy, hormonal therapy, immunotherapy, biological therapy, or radiotherapy within 4 weeks prior to the first study treatment.
* Patient has had major surgery within 4 weeks of the first study treatment.
* Patient has received a blood transfusion, erythropoietin, G-CSF or GM-CSF within 4 weeks.
* Patient has baseline laboratory values that are outside of the normal ranges or those listed (see Inclusion Criteria), which are clinically significant, as determined by the investigator.
* Patient has lost 10% or more of body weight in the previous 3 months.
* Patient has frequent vomiting or severe anorexia.
* Patient has a serious, concurrent medical condition that would limit the patient's ability to complete or comply with the study requirements.
* Patient is unable or unwilling to comply with the contraceptive requirements during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
Efficacy: sum of complete responders and partial responders
Safety: a decrease in cardiac ejection fraction by multigated acquisition (MUGA) scans

SECONDARY OUTCOMES:
Percent of eligible patients with progressive disease (PD)
Percent of patients with stable disease (SD)
Percent of patients with complete response (CR)
Percent of patients with partial response (PR)
Overall response (sum of CR, PR, and SD)
Time to progression (TTP)
Presence and severity of new electrocardiogram (ECG) abnormalities
Presence and severity of myelosuppression (bone marrow suppression)
Presence and severity of alopecia (hair loss)
Presence and severity of stomatitis
Presence and severity of nausea
Presence and severity of vomiting

CONTACTS AND LOCATIONS:
Overall Officials: John H. Ward, MD, Principal Investigator — Hunstman Cancer Institute, University of Utah School of Medicine, Salt Lake City, UT
Locations (3):
- Huntsman Cancer Center, University of Utah, Salt Lake City, Utah, United States
- Bulgaria (2):
  - Sofia Cancer Center, Sofia
  - University Hospital Queen Joanna, Sofia